CLINICAL TRIAL: NCT04675164
Title: Outcome of ICSI Using Laser Assisted Sperm Selection of Viable Immotile Testicular Sperm in Azoospermic Infertile Men: a Randomized Controlled Trial
Brief Title: Laser Assisted Sperm Selection of Viable Immotile Testicular Sperm in Azoospermic Infertile Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Alaa El-Dein Hasan, Assistant Lecturer of Dermatology, Venreology and Andrology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAISS
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Azoospermia; IVF
Keywords: Laser Assisted Immotile Sperm Selection; Hypo-osmotic swelling test; ICSI; Testicular sperm
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Intervention Model Description: (LAISS) group: viable immotile testicular sperms will be selected before ICSI using laser assisted immotile sperm selection (study group).
  (HOST) group: viable immotile testicular sperms will be selected before ICSI using hypo-osmotic swelling test (control group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: With an online tool, participants will be randomized to undergo ICSI with HOST and LAISS sperm selection arms with a 1:1 allocation ratio as per a computer-generated list, using permuted block sizes of 8, and 16, stratified for sites and fresh or cryopreserved sperm. Results of allocation will be in sealed opaque envelopes labeled with unique random codes. Clinicians, embryologists, and participants in all centers will have no access to allocation results. Upon consent, instructors will assign participants to the relevant group. Embryologists who will perform fertilization check and embryo grading will be unaware of the sperm selection method. Women will undergo only day 5 blastocysts transfer. This trial will also conceal the allocation from participants and clinical team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAISS group (Active Comparator): Viable immotile testicular sperms will be selected before ICSI using laser assisted immotile sperm selection (study group).
  Interventions: Device: Laser Assisted Immotile Sperm Selection
- HOST group (Active Comparator): Viable immotile testicular sperms will be selected before ICSI using hypo-osmotic swelling test (control group).
  Interventions: Procedure: Hypo-osmotic Swelling Test

INTERVENTIONS:
Device: Laser Assisted Immotile Sperm Selection — LAISS will be performed using diode laser system at the lowest working power with a single laser shot at the lower one third of the sperm tail. If sperm tail curling occurred, the sperm is then viable and will be utilized for ICSI after immobilization in PVP.
  Arms: LAISS group
Procedure: Hypo-osmotic Swelling Test — HOST will be performed by transferring immotile sperms from incubation droplet into HOST droplet, with any sperm showing tail swelling will be identified as viable and will be utilized for ICSI after immediate transfer and immobilization.
  Arms: HOST group

SUMMARY:
This study aims to investigate the outcome of ICSI after using LAISS for selection of viable immotile testicular sperm in azoospermic infertile men.

Patients will be randomly assigned to 2 groups. In (LAISS) group, viable immotile testicular sperms will be selected before ICSI using laser assisted immotile sperm selection (study group). In (HOST) group, viable immotile testicular sperms will be selected before ICSI using hypo-osmotic swelling test (control group).

ELIGIBILITY:
Inclusion Criteria:

* Eligible couples are those undergoing ICSI due to azoospermia with testicular biopsy positive for sperm (either fresh or cryopreserved) following testicular sperm extraction (TESE) or aspiration (TESA).

Exclusion Criteria:

* Cases with female factor infertility or woman age above 35 years will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6- 7 weeks
  Presence of a fetal heartbeat at 6-7 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan SA Saleh, MD, Study Director — Sohag Faculty of Medicine
Locations (1):
- Ajyal Hospital, IVF Center, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Share IPD upon justified request to study director
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data shall become permanently available for share in Q3 2022.
Access Criteria: Justified request to study director